CLINICAL TRIAL: NCT00727181
Title: An Observational, Prospective Evaluation of the Trifecta™ Valve
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CS05002TV
Record Dates: First submitted 2008-07-29; First posted 2008-08-01 (Estimated); Last update posted 2019-02-04 (Actual); Status verified 2019-02

CONDITIONS: Aortic Valve Insufficiency; Regurgitation, Aortic Valve; Aortic Valve Incompetence; Aortic Valve Stenosis
Keywords: aortic valve; heart valve; tissue valve; bioprosthesis; valve disorder; valve disease; cardiac surgery; aortic valve stenosis; aortic valve regurgitation
MeSH Terms: conditions — Aortic Valve Insufficiency; Aortic Valve Stenosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Trifecta Valve (Other): The Trifecta valve is a tri-leaflet stented pericardial valve designed for supra-annular placement in the aortic position.
  Interventions: Device: Trifecta aortic heart valve

INTERVENTIONS:
Device: Trifecta aortic heart valve — Replacement of a diseased, damaged, or malfunctioning aortic heart valve

SUMMARY:
This trial is designed to confirm the clinical safety and effectiveness of the Trifecta valve by establishing associated adverse event rates, clinical status as indicated by New York Heart Association (NYHA) functional classification, hemodynamic performance, and hematology analysis.

DETAILED DESCRIPTION:
The clinical investigation is a multi-center, multi-country, prospective, non-randomized, observational study without concurrent or matched controls, designed to evaluate the safety and effectiveness of the Trifecta valve. A maximum of 120 subjects requiring aortic valve replacement will be implanted at a maximum of 6 investigational sites in Europe. The sample size is based on late patient-years of follow-up with a minimum of 400 late patient-years experience required.

ELIGIBILITY:
Inclusion Criteria:

1. Patient requires aortic valve replacement. (Note: patients undergoing concomitant procedures, e.g. coronary artery bypass grafting, or valve repair, are eligible for this study).
2. Patient is legal age in host country.
3. Patient (or legal guardian) has given written informed consent for participation prior to surgery.
4. Patient is willing to undergo all study procedures and adhere to data collection and follow-up requirements.

Exclusion Criteria:

1. Patient is pregnant or nursing (women of child bearing potential must have a documented negative pregnancy test within one week prior to surgery).
2. Patient already has a prosthetic valve(s) at a site other than the aortic valve.
3. Patient requires concomitant replacement of the tricuspid, pulmonary, or mitral valve.
4. Patient has an inability or is unwilling to return for the required follow-up visits.
5. Patient has active endocarditis (patients with previous endocarditis must have two documented negative blood culture results prior to enrollment).
6. Patient has had an acute preoperative neurological event defined as patient has not returned to baseline or has not stabilized 30 days prior to the planned valve implantation surgery.
7. Patient is undergoing renal dialysis.
8. Patient has a documented history of substance abuse within one year of enrollment or is currently a prison inmate.
9. Patient is currently participating in the study of an investigational drug or device, or the patient was previously participating in an investigational drug study and has not completed a 30-day wash out period.
10. Patient had the Trifecta valve implanted as part of this study, but then had the device explanted.
11. Preoperative evaluation indicates other significant cardiovascular abnormalities such as aortic dissection or ventricular aneurysm.
12. Patient has a life expectancy less than two years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2007-11; Primary Completion 2010-07 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
To characterize patient NYHA functional classification status | CE labelling
To characterize the hemodynamic performance of the valve, as per echocardiography | CE labelling
Safety outcomes | CE labelling

CONTACTS AND LOCATIONS:
Overall Officials: Friedrich W Mohr, MD, Principal Investigator — Universitat Herzzentrum Leipzig GmbH
Locations (4):
- Hôpital de Pontchaillou, Rennes, France
- Germany (2):
  - Universitat Herzzentrum Leipzig GmbH, Leipzig
  - Deutsches Herzzentrum München, München
- Onze Lieve Vrouwe Gasthuis, Amsterdam, Netherlands